CLINICAL TRIAL: NCT00333450
Title: Multicentre Immune Memory Study in Healthy Children Following a 3 Dose Primary Vaccination With Prevenar or GSK Biologicals' Pneumococcal Conjugate Vaccine Via the Administration of a Single Booster Dose of Pneumovax 23
Brief Title: Immune Memory Evaluation in Children Following a Primary Vaccination With Pneumococcal Conjugate Vaccines.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106623
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Streptococcal
MeSH Terms: conditions — Streptococcal Infections | interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal vaccine

SUMMARY:
To evaluate the immunological memory against pneumococcal vaccine serotypes in children primed with conjugate vaccines by administering a booster dose of plain polysaccharide vaccine.

DETAILED DESCRIPTION:
2 groups (60 per group), booster of Pneumovax 23 after priming with Prevnar or GSK Biologicals' pneumococcal vaccine.

ELIGIBILITY:
Inclusion:

* healthy children between 11-14 months old who received primary vaccination with Prevnar or GSK Biologicals' pneumococcal conjugate vaccine.

Exclusion:

* children having received or planning to receive any investigational products, vaccines not foreseen in the protocol and immune modifying drugs;
* children having received any additional pneumococcal vaccine than in the primary study;
* children with any disease that affect the immune system and history of seizures and/or allergic disease.

Ages: 11 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Antibody concentrations against pneumococcal serotypes 1 month post-booster

SECONDARY OUTCOMES:
Immunogenicity pre and post-booster and safety (follow up of SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- Germany (25):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Marbach, Baden-Wurttemberg
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Tutzing, Bavaria
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Stollberg, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Weimar, Thuringia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Knuf M, Pankow-Culot H, Grunert D, Rapp M, Panzer F, Kollges R, Fanic A, Habib A, Borys D, Dieussaert I, Schuerman L. Induction of immunologic memory following primary vaccination with the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in infants. Pediatr Infect Dis J. 2012 Jan;31(1):e31-6. doi: 10.1097/INF.0b013e3182323ac2. PMID 21909049
- See also: Primary Study — http://www.clinicaltrials.gov/ct/show/NCT00307541
- Available data/document: Statistical Analysis Plan: 106623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register